CLINICAL TRIAL: NCT03980574
Title: Dietary Supplementation in Heart Failure
Acronym: R-DRINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Vascular Scientific, LLC (Unknown)
Responsible Party: Principal Investigator, Sitaramesh Emani, Professor of Medicine, Physiology, and Cell Biology Chair of Excellence in Cardiovascular Medicine Director, Division of Cardiovascular Medicine Deputy Director, Davis Heart and Lung Research Institute, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017H0214
Record Dates: First submitted 2018-08-14; First posted 2019-06-10 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 2 arms of studying with first arm involving a cross-over from active intervention to no intervention and a second arm involving active intervention with no cross-over.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crossover Group (Experimental): The crossover group will be further randomly assigned (1:1) with 20 patients in each group. The two crossover arms of the study will follow the patients for 8 weeks. At the end of week 8, all crossover patients will have a 1 week wash out period. Thereafter, patients will be crossed-over to the opposing arm of the study for an additional 1+8 weeks (R Drink 8 oz 3-5x/day versus a placebo drink 8 oz 3-5x/day).
  Interventions: Dietary Supplement: R Drink
- Non-crossover Group (Experimental): The non-crossover group of the study will follow 20 patients for the entire 17 weeks and participants in this arm will not be crossed over, will not have a washout period, and will consume R Drink for the total duration of the study. If patients in this arm wish to continue on the R Drink, for 6 additional months they may do so. At the end of the optional 6 months these patients will have a repeat research transthoracic echocardiogram. Data collection will occur at baseline, week 8, and week 17. An additional 6 month data collection time point will occur for patients in the third arm opting to continue R Drink.
  Interventions: Dietary Supplement: R Drink

INTERVENTIONS:
Dietary Supplement: R Drink — R Drink is a dietary supplement drink containing filtered reverse osmosis water and 150 mg/L of both USP Grade calcium chloride and magnesium chloride, 10 mg/L Biotin (vitamin B7), 500 mg/L of Niacinamide (B3) and 550 mg/L of Choline.

SUMMARY:
A single-center, double-blind, placebo-controlled, cross-over study pilot study comparing R Drink vs. placebo in 60 heart failure patients. Half of the participants will also have diabetes mellitus. The 60 patients will be distributed among three arms. Total distance walked in six minutes and hospital readmission rates will be examined. Eligible heart failure patients include those with systolic or diastolic heart failure and diabetes mellitus can be Type I or II. All patients will continue on their standard heart failure and diabetes therapies while they participate in the study.

DETAILED DESCRIPTION:
Heart failure (HF) affects millions of Americans, with approximately five-hundred thousand new cases diagnosed annually, with 40% or more of patients having a concomitant diagnosis of diabetes or prediabetes. HF is not a diagnosis itself, but rather a constellation of signs and symptoms due to impaired ventricular filling or ejection of blood. Some of the most common symptoms associated with heart failure include dyspnea, impaired exercise tolerance, and lower extremity edema. Certain co-morbidities like hypertension (HTN) and DM are found more commonly in conjunction with HF. In fact, diabetes is an independent predictor of heart failure. Patients with heart failure and diabetes can have additional clinical symptoms of peripheral neuropathy and poor wound healing, often leading to foot ulcers. The mainstay of treatment for HF at present, employs the use of goal directed medical therapy (GDMT) and cardiac resynchronization therapy (CRT).

Despite these treatments, HF still accounts for over 20% of all hospital admissions in people older than 65. The estimated cost for HF admissions in the US is over $35 billion.

In limited case study, testing participants with a variety of chronic diseases, including HF and DM, observations suggest the incorporation of a dietary supplement drink (R Drink) containing filtered reverse osmosis water and 150 mg/L of both USP Grade calcium chloride and magnesium chloride, 10 mg/L Biotin (vitamin B7), 500 mg/L of Niacinamide (B3) and 550 mg/L of Choline may be beneficial, which is the goal of this unique three-arm clinical trial.

These ingredients are Generally Recognized as Safe (GRAS) ingredients by the FDA and have multiple proposed mechanisms of action which include improved circulation and enhancing clearance of metabolic waste. These electronutrients play a role in the regulation of acetylcholine induced endothelium-dependent relaxation and regulation of nitric oxide, directly influencing vascular tone. They are involved in the s-adenosylmethionine and myelin pathways of the central nervous system, and promote the repair and protection of myelin which is essential for nerve conduction. These electronutrients may promote activation of adenosine triphosphate (ATP) which improves muscular contractions and nerve-muscle impulse transmission. Finally, by regulating the release of serum free fatty acid release, these specific electronutrients may assist in insulin regulation.

This pilot study will be a single center, double-blind, placebo controlled, cross-over study having three arms with a total of 60 patients - all with HF and half with DM - and will compare R Drink versus placebo on the distance walked in 6 minutes, and hospital readmission rates. Eligible patients will have a known diagnosis of HF (diastolic - HFpEF or systolic - HFrEF) classified as NYHA I-IV, a known diagnosis of DM (type I or type II) and will be selected from a larger population being followed in the Heart Failure Clinic at the Ohio State University Wexner Medical Center. All patients will continue on the standard HF and DM therapies as guided by their treating physician. Enrolled patients will be randomly assigned (2:1) to a crossover group (40 patients) and a non-crossover group (20 patients). The crossover group will be further randomly assigned (1:1) with 20 patients in each group. The two crossover arms of the study will follow the patients for 8 weeks. At the end of week 8, all crossover patients will have a 1 week wash out period. Thereafter, patients will be crossed-over to the opposing arm of the study for an additional 1+8 weeks (R Drink 8 oz 3-5x/day versus a placebo drink 8 oz 3-5x/day).

The third arm of the study will follow 20 patients for the entire 17 weeks and participants in this arm will not be crossed over, will not have a washout period, and will consume R Drink for the total duration of the study. If patients in this arm wish to continue on the R Drink, for 6 additional months they may do so. At the end of the optional 6 months these patients will have a repeat research transthoracic echocardiogram. Data collection will occur at baseline, week 8, and week 17. An additional 6 month data collection time point will occur for patients in the third arm opting to continue R Drink.

At the end of study participation, all patients in the two arms that cross will have the study drink discontinued and will continue to follow standard heart failure and diabetic therapies as guided by their treating physicians. The study will use a permuted block randomization. This design should result in a balance of known and unknown con-founders and prevent identification of the randomization sequence, minimizing potential selection bias due to investigator preference. The groups should have the same baseline characteristics and be evenly distributed. Each of the 20 patient cohorts should enroll 10 patients with diabetes within each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Confirmed diagnosis of heart failure (NYHA Class I-IV) (all subjects)
* Confirmed diagnosis of diabetes (type I or II) (only 30 subjects)
* At least 3 months of standard, conventional drug therapy for heart failure, including diuretic dosing. Diuretics can be adjusted during the study per the treating physician within a relatively standard dosing scale. Overall medical therapy should be considered maximally tolerated appropriate therapy by the treating physician.
* Ability to participate in 6-minute walk test
* Literacy and ability to complete neuropathic pain and heart failure quality of life questionnaires
* Signed written consent

Exclusion Criteria:

* Contraindications to the consumption of 1L of purified water per day, when taken into consideration that the average patient with HF is recommended to adhere to a 1.5-2 L fluid restriction per day
* Liver cirrhosis / Prior diagnosis of liver failure
* End-stage renal disease requiring hemo/peritoneal dialysis
* CHF admission requiring diuresis within 14 days prior to enrollment date
* Systolic BP < 100 mmHg or diastolic BP < 60 mmHg (at time of randomization)
* Blood glucose < 70 mg/dl (at time of randomization)
* QRS duration > 130 ms
* QTc duration > 480 ms
* Prior diagnosis of moderate to severe COPD
* Uncontrolled systemic systolic/diastolic hypertension (SBP > 160 mmHg or DBP > 100 mmHg)
* Pregnancy
* History of ventricular tachycardia or SCD
* Refusal to consent/inability to provide signed written consent
* Any condition or abnormality that, at the physician's discretion, would compromise subject safety or data integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Hospital Readmission Rates | Day 119
  Number of total hospital readmissions post-enrollment.

OTHER OUTCOMES:
New York Heart Association Functional Class | Day 0, Day 119
  Additional functional assessment will be made by classifying patients into the appropriate New York Heart Association (NYHA) functional class. NYHA HF classification is a clinical assessment based on reported limitations and symptoms and is assigned by medical professionals performing the assessment. NYHA classification is considered a routine component of HF assessment.
Echocardiographic Measurements | Day 0, Day 56, Day 119
  The echo exam will include the assessment of systolic and diastolic function by recommended techniques (left atrial volume/index, doppler mitral inflow velocities, E/A ratio, tissue doppler of mitral valve, E/e' ratio, IVRT, RVSP, DT, global function/LVEF, left ventricular cavity size, 2D biplane simpson, LV volume/mass). Measurements of these parameters are considered part of a routine clinical echocardiographic exam, but will be completed as part of the research study.
Quality of Life Questionnaires | Day 0, Day 56, Day 119
  Quality of life will be assessed with the Minnesota Living with Heart Failure Questionnaire (MLWFQ), which has been validated as tool to measure quality of life. The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses. Thus, scores may range from 0 (zero) to 105, where a lower score is indicative of a better quality of life.
6-Minute Walk Test | Day 0, Day 56, and Day 119
  The 6-minute walk test (6MWT) is a practical and simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. It measures the distance that a patient can quickly walk on a flat, hard surface over 6 minutes. It importantly evaluates the global responses in multiple systems involved in exercise, such as the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, neuromuscular system and metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity, but since most activities of daily living are performed at submaximal levels of exertion, the 6MW distance may better reflect the functional exercise level for daily physical activities.
Serological Assessment | Day 0, Day 56, and Day 119
  B-natriuretic peptide (BNP) and NT-proBNP are serological markers of HF measured in pg/mL.
Serological Assessment | Day 0, Day 56, and Day 119
  (eGFR) measure in mL/min per 1.73 m2 and creatinine levels. The Estimated glomerular filtration rate is the best test to measure your level of kidney function and determine your stage of kidney disease. A doctor can calculate it from the results of your blood creatinine test measured mg/dL, your age, body size and gender.
Serological Assessment | Day 0, Day 56, and Day 119
  C-reactive protein is a surrogate marker of inflammation measured in mg/L.
Serological Assessment | Day 0, Day 56, and Day 119
  lipid panel measures total cholesterol and triglycerides in mg/dL.
Serological Assessment | Day 0, and Day 119
  Hemoglobin A1c reflects a serum glucose over a 3-month time frame will be measured as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Sitaramesh Emani, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided